CLINICAL TRIAL: NCT00615264
Title: A Phase 3, Multinational, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study To Investigate The Clinical Efficacy And Safety of DiaPep277® in Newly Diagnosed Type 1 Diabetes Patients
Brief Title: Efficacy Study of DiaPep277 in Newly Diagnosed Type 1 Diabetes Patients
Acronym: DIA-AID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Andromeda Biotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 901; ISRCTN55429664
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DiaPep277 (Experimental): DiaPep277 1.0 mg + 40 mg Mannitol in 0.5 mL lipid emulsion.
  Interventions: Drug: DiaPep277
- Placebo (Placebo Comparator): Mannitol 40 mg in 0.5 mL lipid emulsion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DiaPep277 — 1.0mg dose, administered as subcutaneous injection, on 0, 1, 3, 6, 9, 12, 15, 18 and 21 months
  Arms: DiaPep277
Drug: Placebo — Mannitol (excipient) 40 mg, administered as subcutaneous injection on 1, 3, 6, 9, 12, 15, 18 and 21 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if DiaPep277 can effectively protect the internal production of insulin in patients newly diagnosed with type 1 diabetes, by stopping the immune destruction of insulin-producing beta-cells in the pancreas. DiaPep277 acts on the immune system and is expected to prevent further destruction of the beta-cells by stimulating regulatory responses, without causing immunological suppression.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 1 diabetes for up to 3 months at screening
* Insulin dependency
* Fasting C-peptide levels >= 0.22 nmol/L
* Presence of at least 1 of the diabetes-related autoantibodies (IA-2A, GAD or IA)

Exclusion Criteria:

* Pregnancy or intent to conceive in the next 2 years
* Significant diseases that could affect response to treatment, such as tumors, psychiatric disorders, substance abuse, severe allergies or diabetes-related complications.
* Patient has immune deficiency or receives immuno-suppressive or cytotoxic drugs.

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 457 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, MD, Principal Investigator — Hadassah Medical Center, Jerusalem; Paolo Pozzilli, MD, Principal Investigator — Universita Campus Bio-Medico, Rome; Francois Bonici, MD, Principal Investigator — New Groote Schuur Hospital, Cape Town; Thomas Linn, MD, Principal Investigator — Universitätsklinikum, Giessen
Locations (34):
- Rudolfstiftung Hospital, Vienna, Austria
- Czechia (3):
  - Faculty Hospital, Olomouc
  - Faculty hospital Motol., Prague
  - IKEM/Diabetes Centre, Prague
- Finland (3):
  - Pohjois-Karjala projektin tutkimussäätiö, Joensuu
  - Tutkimusyksikkö Oulu, Oulu
  - Diabetestutkimus, Vantaa
- France (4):
  - CHU de Grenoble, Grenoble
  - Hopital Edouard Herriot, Lyon
  - Hopital La Timone, Marseille
  - CHU de Nîmes/ Hôpital Caremeau, Nîmes
- Germany (3):
  - Universitätsklinikum, Giessen
  - Diabetes Centre for Children and Adolescents, Hanover
  - Institut für Diabetesforschung an der Klinik und Hochschulambulanz für Kinder- und Jugendmedizin, Munich
- Laiko hospital, Athens, Greece
- Israel (3):
  - Wolfson Medical Centre, Holon
  - Hadassah University Hospital, Jerusalem
  - Schneider Children's Medical Centre, Petah Tikva
- Italy (5):
  - Universita' degli Studi di Bari, Bari
  - Ex Istituto di clinica medica, Palermo
  - University Campus Bio-Medico, Rome
  - Università "La Sapienza", Rome
  - Istituto Clinico Humanitas, Rozzano
- South Africa (5):
  - Helderberg Clinical Trials Unit, Cape Town
  - New Groote Schuur Hospital, Cape Town
  - 102 Parklands Medical Centre, Durban
  - Donald Gordon Medical Center, Johannesburg
  - Centre for Diabetes and Endocrinology, Johannesburg
- Spain (4):
  - Hospital de la Santa Creu, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital de Sabadell, Sabadell
  - Hospital Nuestra Señora de La Candelaria, Santa Cruz de Tenerife
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - Royal Shrewsbury Hospital, Shrewsbury

REFERENCES:
- [Derived] Raz I, Ziegler AG, Linn T, Schernthaner G, Bonnici F, Distiller LA, Giordano C, Giorgino F, de Vries L, Mauricio D, Prochazka V, Wainstein J, Elias D, Avron A, Tamir M, Eren R, Peled D, Dagan S, Cohen IR, Pozzilli P; DIA-AID 1 Writing Group. Treatment of recent-onset type 1 diabetic patients with DiaPep277: results of a double-blind, placebo-controlled, randomized phase 3 trial. Diabetes Care. 2014;37(5):1392-400. doi: 10.2337/dc13-1391. PMID 24757230 (Retraction: PMID 25538317 Diabetes Care. 2015 Jan;38(1):178)
- [Derived] Pozzilli P, Raz I, Peled D, Elias D, Avron A, Tamir M, Eren R, Dagan S, Cohen IR. Evaluation of long-term treatment effect in a type 1 diabetes intervention trial: differences after stimulation with glucagon or a mixed meal. Diabetes Care. 2014;37(5):1384-91. doi: 10.2337/dc13-1392. Epub 2014 Jan 9. PMID 24408401 (Retraction: PMID 25538318 Diabetes Care. 2015 Jan;38(1):179)

RESULTS

PARTICIPANT FLOW:
Groups:
- DiaPep277: DiaPep277 1.0 mg + 40 mg Mannitol in 0.5 mL lipid emulsion.
  DiaPep277: 1.0 mg dose, administered as subcutaneous injection, on 0, 1, 3, 6, 9, 12, 15, 18 and 21 months
Period: Overall Study
Arm/Group | DiaPep277 | Placebo
Started | 225 | 232
Received at Least One Dose (ITT) | 225 | 231
ITT Patients Who Met Inc/Excl (MITT) | 209 | 213
Completed | 175 | 180
Not Completed | 50 | 52
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Lost to Follow-up | 6 | 13
Not completed — Adverse Event | 8 | 5
Not completed — Death | 1 | 1
Not completed — Protocol Violation | 11 | 7
Not completed — Not defined | 7 | 4
Not completed — Dermal Hypersensitivity | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- DiaPep277: DiaPep277 1.0 mg + 40 mg Mannitol in 0.5mL Lipid emulsion.
  DiaPep277: 1.0 mg dose, administered as subcutaneous injection, on 0, 1, 3, 6, 9, 12, 15, 18 and 21 months
- Total: Total of all reporting groups
Arm/Group | DiaPep277 | Placebo | Total
Number analyzed (Participants) | 225 | 231 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.6 (7.99) | 26.4 (7.85) | 26.5 (7.91)
Age, Customized [Median (Full Range); unit: years] | 25.0 [15 to 46] | 26.0 [15 to 46] | 25.0 [15 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 73 | 156
  Male | 142 | 158 | 300
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 212 | 212 | 424
  Black | 6 | 7 | 13
  Oriental | 2 | 1 | 3
  Asian | 1 | 4 | 5
  Other | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glucagon-stimulated C-peptide AUC at 24 Months
Description: Beta-cell function, measured as change in stimulated C-peptide secretion measured 0, 2, 6, 10 and 20 minutes post administration [area under the curve (AUC), 0-20 minutes] at Baseline and 24 months, during a glucagon stimulation test (GST). The change in AUC was calculated per patient by subtracting the baseline AUC from the 24 month AUC.
Time Frame: Baseline and 24 months
Population: Modified Intent to Treat (MITT) Population - all randomized patients who received at least one dose of study medication and who entered the study according to the definition of the target population, as defined by the inclusion and exclusion criteria in the study protocol
Measure: Mean (Standard Error); unit: nmol*minute/L
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 209 | 213
nmol*minute/L | -3.848 (0.4666) | -4.348 (0.4584)
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; Test type: Superiority or Other; p = 0.2851, Mixed Models Analysis; Calculated with terms for treatment, visit, treatment by visit interaction, baseline C-peptide and country with the unstructured option for the matrix

2. Secondary Outcome: Change From Baseline in Mixed-meal Stimulated C-peptide AUC at 24 Months
Description: Beta cell function, measured as stimulated C-peptide secretion from 0 to 120 min post administration AUC, at baseline and 24 month measurements in a mixed-meal tolerance test (MMTT). The change in AUC was calculated per patient by subtracting the baseline AUC from the 24 month AUC.
Time Frame: Baseline and 24 Months
Population: Modified Intent to Treat (MITT) Population
Measure: Mean (Standard Error); unit: nmol*minute/L
Arm/Group | DiaPep277 | Placebo
Number analyzed (Participants) | 209 | 213
nmol*minute/L | -44.33 (3.6884) | -43.24 (3.5898)
Statistical Analysis 1: Comparison: DiaPep277 vs Placebo; Test type: Superiority or Other; p = 0.7690, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: AE data were collected from the time of subject enrollment through three months after the final product administrations (Total of 24 months after first study product administration)
Arm/Group | DiaPep277 | Placebo
Serious Adverse Events (participants affected / at risk) | 26/225 | 14/231
Other Adverse Events (participants affected / at risk) | 173/225 | 164/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DiaPep277 (N=225) | Placebo (N=231)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 4 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2
Accidental Overdose (Psychiatric disorders) | 1 | 1
Hypoglycemic Coma (Metabolism and nutrition disorders) | 1 | 1
Major Depression (Psychiatric disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Alcohol Poisoning (Psychiatric disorders) | 1 | 0
Jaw Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Concussion (Nervous system disorders) | 0 | 1
Head Injury (Nervous system disorders) | 0 | 1
Ligament Rupture (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchopneumomnia (Infections and infestations) | 1 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Gastritis Viral (Gastrointestinal disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Facial Paresis (Nervous system disorders) | 1 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria Cholinergic (Skin and subcutaneous tissue disorders) | 0 | 1
Death (Social circumstances) | 1 | 0 — This patient had an unspecified event leading to their death. The Investigator confirmed that the death certificate and autopsy results were unobtainable.
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Death (Social circumstances) | 0 | 1 — In the placebo group a male patient's wife became pregnant with twins. Both were live births, but one died shortly after due to an intracranial hemorrhage, which was reported in the database within the placebo group
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DiaPep277 (N=225) | Placebo (N=231)
Nasopharyngitis (Infections and infestations) | 37 | 41
Influenza (Infections and infestations) | 30 | 23
Upper respiratory Tract Infection (Infections and infestations) | 23 | 19
Gastroenteritis (Infections and infestations) | 14 | 17
Pharyngitis (Infections and infestations) | 8 | 7
Tonsillitis (Infections and infestations) | 7 | 6
Urinary Tract Infection (Infections and infestations) | 6 | 9
Bronchitis (Infections and infestations) | 6 | 8
Sinusitis (Infections and infestations) | 6 | 8
Cystitis (Infections and infestations) | 6 | 1
Respiratory Tract Infection (Infections and infestations) | 5 | 6
Nausea (Gastrointestinal disorders) | 8 | 6
Gastritis (Gastrointestinal disorders) | 8 | 3
Toothache (Gastrointestinal disorders) | 7 | 3
Diarrhea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 5 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 5
Pyrexia (General disorders) | 10 | 11
Injection Site Erythema (General disorders) | 9 | 3
Injection Site Pain (General disorders) | 8 | 8
Injection Site Induration (General disorders) | 5 | 3
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 28 | 19
Blood Creatine Phosphokinase Increased (Investigations) | 6 | 9
Alanine Aminotransferase Increased (Investigations) | 5 | 3
Glycosylated Haemoglobin Increased (Investigations) | 3 | 7
Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 26 | 21
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Headache (Nervous system disorders) | 12 | 12
Dizziness (Nervous system disorders) | 5 | 1
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Hypercholesterolemia (Metabolism and nutrition disorders) | 2 | 7
Renal and Urinary Disorders (Renal and urinary disorders) | 10 | 4
Reproductive System and Breast Disorders (Reproductive system and breast disorders) | 8 | 7
Psychiatric disorders (Psychiatric disorders) | 8 | 6
Endocrine Disorders (Endocrine disorders) | 7 | 2
Eye Disorders (Eye disorders) | 6 | 5
Anemia (Blood and lymphatic system disorders) | 2 | 5
Hypertension (Vascular disorders) | 3 | 6
Immune System Disorders (Immune system disorders) | 3 | 6
Cardiac Disorders (Cardiac disorders) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall submit any paper or presentation to the Sponsor for review and comments at least 60 days prior to submitting the same to a third party. Upon receiving any request from the Sponsor to delete any Confidential Information or request to delay in publication up to 90 days to allow the filing of any Sponsor application, the Investigator shall take the request action. Investigator shall not be restricted after 18 months from completion of their site's performance in the study.